CLINICAL TRIAL: NCT03374527
Title: Recirculating Memory T Cells in the Pathogenesis of Psoriatic Arthritis and Cutaneous Psoriasis
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: T-ART
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Psoriasis; Psoriatic Arthritis
Keywords: T-cells; circulation; synovial fluid; psoriasis; psoriatic arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells, blood serum, synovial fluid mononuclear cells, synovial fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Psoriasis: Patients with psoriasis vulgarism without clinical signs of PsA
  Interventions: Other: blood sample collection
- Psoriatic Arthritis (PsA): Patients with a diagnosis of psoriatic arthritis and cutaneous psoriasis
  Interventions: Other: blood sample collection; Procedure: Synovial Fluid collection
- Control group: Healthy subjects
  Interventions: Other: blood sample collection

INTERVENTIONS:
Other: blood sample collection — Blood samples are collected from patients with psoriasis vulgaris and patients with psoriatic arthritis following the routine procedure. Blood samples will also be collected from healthy control subjects.
Procedure: Synovial Fluid collection — Synovial fluid is collected when prescribed in patients with psoriatic arthritis
  Groups: Psoriatic Arthritis (PsA)

SUMMARY:
The aim of the study is to investigate the link between pro-inflammatory T cells responses arising in the skin in patients with cutaneous psoriasis and those present in the joints of patients developing psoriatic arthritis.

The study is based on the hypothesis that a fraction of T cells with memory phenotype can recirculate from the skin and relocalize at extracutaneous sites including enthesis or synovial tissue thus propagating the pro-inflammatory cycle. This could represent a pathogenic mechanism in the development of PsA.

The main aim of the study is to define the phenotypic and functional differences of circulating T cells in patients cutaneous psoriasis, patients with psoriatic arthritis and in control group of healthy subject.

To this end the investigators analyze the expression of cell surface markers of central memory (TCM), effector memory (TEM) and effector (Teff) cells, within this subsets the investigators evaluate the expression of chemokine receptors as well as skin and tissue homing molecules. There will be also an evaluation of the T cell polarization towards Th1/Tc1 or Th17/Tc17 phenotype by evaluating the cytokine expression profile.

In selected patients with PsA the researchers analyze in parallel the phenotype and the cytokine profile of T cell subpopulations in peripheral blood and in synovial fluid, The results of this study could possibly allow to define distinctive features of circulating T cells in patients with PsA and to understand the link between circulating and synovial fluid T cells in patients with PsA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cutaneous psoriasis without clinical signs of PsA,
* Patients with a diagnosis of PsA
* Healthy subjects with a negative family and personal anamnesis for psoriasis.
* Absence of acute and chronic systemic or cutaneous infections during sample collections.

Exclusion Criteria:

* Treatment with cyclosporin A, methotrexate, systemic corticosteroids or any other immunosuppressant agent within 3 weeks before the blood samples collections.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of the percentage of different subsets of memory T cells in the circulation of patients with psoriasis, patients with psoriatic arthritis and a control group of healthy subject. | At time of blood collection
  Central memory, Effector memory and Effector cell markers are evaluated in circulating CD4 and CD8 T cells. Within these subsets the expression of chemokine receptors is also evaluated and we define the cytokine secretion profile for each subset.

SECONDARY OUTCOMES:
Correlation between the circulating percentage of individual subsets of CD4 and CD8 T cells and the clinical disease parameters: Psoriasis Area and Severity Index (PASI) Score and serum level of C reactive protein (CRP) | At time of blood collection
  For each subsets it is calculated the correlation between the percentage in the circulation and either the Psoriasis Area and Severity Index (PASI) score or the serum level of C reactive protein
Parallel analysis of the phenotype of CD4 and CD8 T cells in the circulation and in synovial fluid of patients with psoriatic arthritis. | At time of blood and synovial fluid collection
  Phenotype and functional analysis of T Cells

CONTACTS AND LOCATIONS:
Overall Officials: Eva Reali, Dr., Principal Investigator — I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio
Locations (1):
- IRCCS Galeazzi Orthopedic Hospital, Milan, Italy

REFERENCES:
- [Result] Diani M, Galasso M, Cozzi C, Sgambelluri F, Altomare A, Cigni C, Frigerio E, Drago L, Volinia S, Granucci F, Altomare G, Reali E. Blood to skin recirculation of CD4+ memory T cells associates with cutaneous and systemic manifestations of psoriatic disease. Clin Immunol. 2017 Jul;180:84-94. doi: 10.1016/j.clim.2017.04.001. Epub 2017 Apr 6. PMID 28392462
- [Result] Sgambelluri F, Diani M, Altomare A, Frigerio E, Drago L, Granucci F, Banfi G, Altomare G, Reali E. A role for CCR5(+)CD4 T cells in cutaneous psoriasis and for CD103(+) CCR4(+) CD8 Teff cells in the associated systemic inflammation. J Autoimmun. 2016 Jun;70:80-90. doi: 10.1016/j.jaut.2016.03.019. Epub 2016 Apr 8. PMID 27068801
- [Derived] Casciano F, Diani M, Altomare A, Granucci F, Secchiero P, Banfi G, Reali E. CCR4+ Skin-Tropic Phenotype as a Feature of Central Memory CD8+ T Cells in Healthy Subjects and Psoriasis Patients. Front Immunol. 2020 Apr 3;11:529. doi: 10.3389/fimmu.2020.00529. eCollection 2020. PMID 32318062